CLINICAL TRIAL: NCT05190575
Title: An Open-label, Single-arm Phase II Study to Evaluate the Efficacy and Safety of TST001 for Patients With CLDN18.2 Positive Previously Treated Unresectable Advanced or Metastatic Biliary Tract Cancer
Brief Title: TST001 in Patients With CLDN18.2 Positive Previously Treated Advanced Biliary Tract Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Collaborators: Transcenta Holding Limited (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTC-II-CLDN18.2-TST001
Record Dates: First submitted 2021-12-28; First posted 2022-01-13 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2021-12

CONDITIONS: Biliary Tract Neoplasms
MeSH Terms: conditions — Biliary Tract Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TST001 (Experimental): Drug: TST001 IV infusion every 3 weeks until disease progression or other discontinuation criteria.
  Interventions: Drug: TST001

INTERVENTIONS:
Drug: TST001 — TST001 IV infusion every 3 weeks until disease progression or other discontinuation criteria.

SUMMARY:
TST001 is a recombinant humanized anti-Claudin 18.2 (CLDN18.2) IgG1 monoclonal antibody. This is an open-label, single-arm phase II study to evaluate the efficacy and safety of TST001 for patients with CLDN18.2 positive previously treated unresectable advanced or metastatic Biliary Tract Cancer.

DETAILED DESCRIPTION:
TST001 is a recombinant humanized anti-Claudin 18.2 (CLDN18.2) IgG1 monoclonal antibody. Claudin18.2 (CLDN18.2) protein is one of the family of tetraspanning proteins expressed at epithelial tight junctions and primarily expressed only in normal gastric tissues . CLDN18.2 protein is a pancancer target expressed in primary lesions and metastases of variouscancer types, including gastric cancer, biliary tract cancer and others. Current available information indicates that CLDN18.2 is a promising therapeutic target for the treatment of solid tumors.

This is an open-label, single-arm phase II study to evaluate the efficacy and safety of TST001 for patients with CLDN18.2 positive previously treated unresectable advanced or metastatic Biliary Tract Cancer. Eligible patients will be treated with TST001 until disease progression or other discontinuation criteria met. If there is ≥ one objective response among the first 15 enrolled patients, then the trial continues to enroll a total of 40 patients; if not, then the trial discontinues.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, unresectable advanced or metastatic biliary tract cancer.
* Patients failed at least one prior line of systemic medications; if patients had disease progression during or within 6 months after the completion of adjuvant therapy or neoadjuvant therapy, the adjuvant therapy or neoadjuvant therapy could be regarded as one line of therapy.
* CLDN18.2 expression positive confirmed through tumor tissue.
* Patients with at least one measurable disease according to RECISTv1.1.
* ECOG PS of 0 or 1.
* Patients have predicted life expectancy ≥ 12 weeks.
* Paitients with adequate cardica, liver, renal function, etc.

Exclusion Criteria:

* • History of another concurrent primary malignancy.

  * Untreated or symptomatic CNS metastases.
  * Prior treatment targeting CLDN18.2.
  * Major surgical procedure, prior locoregional therapy such as radioembolization within 28 days prior to the first dose of study drug.
  * Prior serious hypersensitivity to monoclonal antibody or any component of the investigational drug.
  * Patients had any of the following within 6 months prior to first dose of study treatment: cerebrovascular accident, transient ischemic attack, myocardial infarction or unstable angina pectoris, heart failure NYHA III or IV degree, or uncontolled uarrhythmia requiring intervention.
  * Patients who are pregnant or lactating.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2023-05-06 (Actual); Study Completion 2023-05-06 (Actual)

PRIMARY OUTCOMES:
ORR | 18 months
  ORR according to RECIST 1.1 using investigator assessment

SECONDARY OUTCOMES:
PFS | 18 months
  PFS accorridng RECSIST1.1 using investigator assessment
Overall survival | 18 months
  Time from enrollment to death of any cause
DoR | 18 months
  DoR accroding to RECSIST1.1 using investigator assessment
DCR | 18 months
  Patients who were assessed as partial response, complete response or stable disease
Safety & tolerability | 18 months
  Adverse events will be graded according to NCI-CTC AE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Jia Fan, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- Zhongshan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No